CLINICAL TRIAL: NCT04312165
Title: DuraMesh Laparotomy Closure Following Trauma and Emergency Surgery: A Prospective Clinical Trial to Evaluate the Safety and Efficacy of DuraMesh Laparotomy Closure Following Trauma or Emergency Surgery and for Delayed Primary Closure of the Abdomen
Brief Title: DuraMesh Laparotomy Closure Following Trauma and Emergency Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Financial
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gregory Dumanian, LCDR, Staff Surgeon Plastic and Reconstructive Surgery, Uniformed Services University of the Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00083440
Record Dates: First submitted 2020-03-08; First posted 2020-03-18 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Hernia Incisional; Suture, Complication
Keywords: mesh; suture; laparotomy; incisional hernia; prevention
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Intervention Model Description: 2:1 randomization between Duramesh closure and standard suture closure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Duramesh Laparotomy Closure (Experimental): Patients undergoing a midline laparotomy for trauma or emergency surgery will be randomized to either #1 Duramesh suture or standard suture, which is a #1 slowly-absorbing PDS single strand or looped suture based on surgeon preference.
  Interventions: Device: Duramesh Laparotomy Closure
- Control group-Conventional suture closure (Active Comparator): Patients undergoing a midline laparotomy for trauma or emergency surgery will be randomized to either #1 Duramesh suture or standard suture, which is a #1 slowly-absorbing PDS single strand or looped suture based on surgeon preference.
  Interventions: Device: Conventional suture closure

INTERVENTIONS:
Device: Duramesh Laparotomy Closure — Closure of midline laparotomy incision with experimental suture
  Other Names: mesh suture
  Arms: Duramesh Laparotomy Closure
Device: Conventional suture closure — Closure of midline laparotomy incision with standard suture
  Other Names: polydiaxanone; PDS
  Arms: Control group-Conventional suture closure

SUMMARY:
The proposed project aims to evaluate the safety of DuraMesh™ suture for laparotomy closure in an emergent setting, while also providing preliminary efficacy data with regard to incisional hernia prevention. Conventional techniques for laparotomy closure in the setting of an emergency laparotomy or delayed abdominal closure suffer from a lack of durability, with incisional hernia rates of 30-34% reported. While prophylactic planar mesh placement has emerged as a cost-effective strategy to prevent hernia formation in the clean, elective laparotomy setting, higher rates of surgical site complications and increased technical complexity preclude its use in the emergency or contaminated setting. Utilized exactly like conventional suture without any change in surgical closure technique, DuraMesh™ provides the durability of planar mesh reinforcement without the marked increase in foreign material or added surgical complexity. As a result, DuraMesh™ is the only hernia prevention strategy that can be forward-deployed in support of the injured warfighter. While this study is specifically targeted to a gap in the care of the injured warfighter, the potential benefits extend well beyond the military applications. With over 2 million laparotomies performed annually in the United States, and approximately 20% of these resulting in an incisional hernia, the need for an alternative abdominal wall closure strategy is equally dire in the civilian setting. This clinical trial represents an opportunity to drive the needed paradigm shift towards prevention, rather than costly management of incisional hernias. The investigators anticipate this work will rapidly lead to further research, including providing the preliminary data necessary to launch a multi-center randomized controlled trial to assess the clinical efficacy of DuraMesh™ for hernia prevention in both the emergent and elective operative settings.

DETAILED DESCRIPTION:
This is a multisite randomized control proof-of-concept trial to evaluate the safety of DuraMesh™ laparotomy closure in the trauma and emergency laparotomy setting. Approximately 120 patients will be randomized (2:1) to DuraMesh™ laparotomy closure versus conventional suture closure. #1 DuraMesh™ will be provided for patients assigned to the DuraMesh™ treatment arm. Patients will participate in a one-year follow-up regime (2 weeks,1 month, 3 months, 6 months and 12 months).

Primary Laparotomy Closure Treatment 1) Study Group - DuraMesh™ Laparotomy Closure (DLC) Treatment 2) Control Group - Conventional Suture Closure (CSC)

Patients undergoing a midline laparotomy for trauma or emergency surgery will be randomized to either #1 DuraMesh™ suture or conventional laparotomy closure using size #1 slowly-absorbing (PDS) single strand or looped suture, based on surgeon preference. All patients will be assessed for post-operative complications at 2 weeks, 1 month, 3 months, 6 months, and 12 months postoperatively. Patients will also be assessed for incisional hernia formation at the same post-operative time points (2 weeks,1 month, 3 months, 6 months, 12 months). Hernia outcomes will be based on physical examination, with ultrasound used for any uncertainties.

ELIGIBILITY:
Inclusion Criteria:

* Midline laparotomy 5 cm (2 inches) long
* Urgent or emergent surgery following trauma
* Urgent or emergent surgery for diverticulitis
* Urgent or emergent surgery for large or small bowel obstruction
* Urgent or emergent surgery for exploratory laparotomy for acute abdomen
* Urgent or emergent surgery for exploratory laparotomy for intraabdominal hemorrhage

Exclusion criteria

* Inability to provide informed consent
* Prior Hernia repair or existing ventral hernia mesh EXCLUDING inguinal hernias
* Metastatic cancer
* Pregnancy
* Immunosuppression

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Rate of surgical site infection | 30 days
  hematoma, seroma, dehiscence, fistula, bowel obstruction, removal infected mesh suture, return to OR, readmission, mortality

SECONDARY OUTCOMES:
Intraoperative endpoints | day zero, time of implantation
  length of surgery procedure, length of hospital stay, length of laparotomy incision
Rate of incisional hernia formation | within 12 months
  clinical or radiographic evidence of hernia formation
Quality of life patient reported outcomes | 1 month
  SF-36 questionnaire, Scale 0-100, 100 implies no disability
Quality of life patient reported outcomes | 3 month
  SF-36 questionnaire, Scale 0-100, 100 implies no disability
Quality of life patient reported outcomes | 6 months
  SF-36 questionnaire, Scale 0-100, 100 implies no disability
Quality of life patient reported outcomes | 12 months
  SF-36 questionnaire, Scale 0-100, 100 implies no disability
Abdominal wall function patient reported outcomes | 1 month
  HerQles patient reported outcomes for abdominal wall function, Scale 0-100, 100 implies excellent abdominal wall function
Abdominal wall function patient reported outcomes | 3 months
  HerQles patient reported outcomes for abdominal wall function, Scale 0-100, 100 implies excellent abdominal wall function
Abdominal wall function patient reported outcomes | 6 months
  HerQles patient reported outcomes for abdominal wall function, Scale 0-100, 100 implies excellent abdominal wall function
Abdominal wall function patient reported outcomes | 12 months
  HerQles patient reported outcomes for abdominal wall function, Scale 0-100, 100 implies excellent abdominal wall function
Pain patient reported outcome | 1 month
  Numerical pain rating scale, Scale 0-10, 0 implies no pain
Pain patient reported outcome | 3 months
  Numerical pain rating scale, Scale 0-10, 0 implies no pain
Pain patient reported outcome | 6 months
  Numerical pain rating scale, Scale 0-10, 0 implies no pain
Pain patient reported outcome | 12 months
  Numerical pain rating scale, Scale 0-10, 0 implies no pain
Visual analog scale pain, patient reported outcome | 1 month
  Wong-Baker faces pain scale, Scale 0-10, 0 implies no pain
Visual analog scale pain, patient reported outcome | 3 months
  Wong-Baker faces pain scale, Scale 0-10, 0 implies no pain
Visual analog scale pain, patient reported outcome | 6 months
  Wong-Baker faces pain scale, Scale 0-10, 0 implies no pain
Visual analog scale pain, patient reported outcome | 12 months
  Wong-Baker faces pain scale, Scale 0-10, 0 implies no pain

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Maryland Shock Trauma, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Undecided